CLINICAL TRIAL: NCT04085263
Title: The Effect of Rhomboid Intercostal and Subserratus Plane Block on the Postoperative Analgesia of Patients Undergoing Radical Mastectomy: Randomized Controlled Study
Brief Title: Rhomboid Intercostal and Subserratus Plane Block
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Tanta University (Other)
Collaborators: Dr. Mohamed shebl Abdelghany (Unknown)
Responsible Party: Principal Investigator, Sameh Abdelkhalik Ahmed Ismaiel, Dr, Tanta University
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Supportive Care
Other Study IDs: 33206/07/19
Record Dates: First submitted 2019-09-09; First posted 2019-09-11 (Actual); Last update posted 2022-09-13 (Actual); Status verified 2022-09

CONDITIONS: Postoperative Pain; Regional Anesthesia Morbidity
Keywords: Radical Mastectomy; Postoperative pain; Morphine consumption; subserratus plane block
MeSH Terms: conditions — Pain, Postoperative | interventions — Control Groups

STUDY DESIGN:
Intervention Model Description: Prospective study
Who Masked: Participant, Investigator, Outcomes Assessor
Masking Description: The participants will be kept blind through the use of sham block in the control group.
  Outcome assessors will be blinded as they will be anesthesia resident and nurse not participating in the study.
  The investigators will be blinded
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Control group (Sham Comparator): The patients in this group will receive sham rhomboid intercostal and subserratus plane.
  Interventions: Procedure: Control group
- Rhomboid intercostal and subserratus plane block group (Experimental): The patients in this group will be receive real ultrasound-guided rhomboid intercostal and subserratus plane.
  Interventions: Procedure: Rhomboid intercostal and subserratus plane block group

INTERVENTIONS:
Procedure: Control group — The patients in this group will receive sham rhomboid intercostal and subserratus plane.
  Other Names: Sham block group
  Arms: Control group
Procedure: Rhomboid intercostal and subserratus plane block group — The patients in this group will be receive real ultrasound-guided rhomboid intercostal and subserratus plane.
  Other Names: Experimental group
  Arms: Rhomboid intercostal and subserratus plane block group

SUMMARY:
This clinical trial will be conducted at Tanta University Hospitals, General Surgery Hospitals on female patients undergoing radical mastectomy

. All the patients will receive general anesthesia.

The patients will be randomly allocated into one of the following two groups;- - Control group (30 patients): The patients in this group will receive sham rhomboid intercostal and subserratus plane.

- Rhomboid intercostal and subserratus plane block group (30 patients): The patients in this group will be receive real ultrasound-guided rhomboid intercostal and subserratus plane.

The primary outcome measure will be the total dose of morphine consumed in the first 24 h after surgery and the secondary outcome will be the postoperative pain score.

DETAILED DESCRIPTION:
This prospective randomized controlled study will be carried out on female patients who will be presented for radical mastectomy in the general surgery department in Tanta university hospitals over three month duration and 6 months follow up that starts immediately after obtaining ethical committee approval, an informed written consent will be obtained from all the participants, all patients data will be confidential and will be used for the current study only.

Any unexpected risks that will appear during the research will be announced to the participants and to the ethical committee at time and adequate measures will be taken to resolve and avoid these risks.

Expected risks to the patients: patients enrolled in this study will minimal risk of local hematoma that which will be managed by adequate compression and minimal risk of infection that will be guarded against by adequate sterilization and prophylactic antibiotic.

There will be adequate supervision to maintain the privacy of patients and confidentiality of data.

There will be no conflict of interest, nor conflict with religion, law, or society standards.

The research will be beneficial to the society and has no risk of environmental pollution.

Upon arrival of the patient to the operating room, intravascular access will be established, fluid preload will be started, and basic monitor will be attached. After positioning and adequate sterilization of the back. The patients will be randomly allocated into two equal groups by the aid of computer-generated software of randomization; - • Control group (30 patients): The patients in this group will receive sham rhomboid intercostal and subserratus plane.

• Rhomboid intercostal and subserratus plane block group (30 patients): The patients in this group will be receive real ultrasound-guided rhomboid intercostal and subserratus plane.

Anesthesia will be induced by fentanyl 1 ug/kg, propofol 1.5 mg/kg, and cis-atracurium 0.15 mg/kg to facilitate tracheal intubation. After endotracheal intubation, the patients will be connected to a mechanical ventilator with its parameters adjusted to maintain etCo2 32-36 mmhg. Anesthesia will be maintained by isoflurane 1% MAC in mixture of oxygen:air 1:1 with the use of low flow (1 ml/min).

All the patients will be connected to a bispectral index monitor with maintaining its value ranging 40-60. Increase in the BIS value over 60 will be managed by additional dose of fentanyl 1ug/kg till decrease the BIS below 60. If the BIS is still over 60, increasing the isoflurane 0.2 % MAC till it decreased below 60.

At the end of the surgery, switching off the inhalational anesthetics, reversal of muscle relaxation, and awake tracheal extubation will be done with transporting the patients to the PACU for postoperative follow up and monitoring.

ELIGIBILITY:
Inclusion Criteria:

* Female patients
* Aged 40-75 years
* ASA class I-II
* Presented for elective radical mastectomy.

Exclusion Criteria:

* Patients refused to participate.
* Patients with known or suspected allergy to the used medication.
* Patients with preoperative chronic pain
* Patients received preoperative opioids or gabapentoids.
* Patients with major cardiac, renal, respiratory, or hepatic disease.
* Patients with potential risk of coagulopathy
* Uncooperative patients.
* Obese patients with BMI >36

Ages: 40 Years to 75 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 69 (Actual)
Dates: Start 2019-09-01 (Actual); Primary Completion 2022-09-06 (Actual); Study Completion 2022-09-06 (Actual)

PRIMARY OUTCOMES:
The postoperative morphine consumprtion | The first 24 hours postoperatively
  3 mg morphine i.v will be given when the postoperative VAS score was 4 or more considering the total dose consumption in the first postoperative day not exceeding 15 mg

SECONDARY OUTCOMES:
The postoperative pain score | The first 24 hours postoperatively
  The postoperative Visual analogue score

CONTACTS AND LOCATIONS:
Overall Officials: Sameh Ismaiel, M.D, Principal Investigator — Lecturer of Anesthesia and Intensive Care, Tanta University
Locations (1):
- Tanta University hospitals, Tanta, Egypt

IPD SHARING:
Plan to Share IPD: No
Once the study had been successfully completed, the data will be shared for other researchers.